CLINICAL TRIAL: NCT02777021
Title: Home or Away From Home: Comparing Patient and Caregiver Reported Quality of Life (QoL) and Other Patient-centered Outcomes for Inpatient Versus Outpatient Management of Neutropenia in Children With AML
Brief Title: Home Away From Home - Quality of Life Surveys
Acronym: Aim 3
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Healthcare of Atlanta (Other); C.S. Mott Children's Hospital (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Arkansas Children's Hospital Research Institute (Other); Children's Medical Center Dallas (Other); Baylor College of Medicine (Other); Primary Children's Hospital (Other); Children's Hospital of Michigan (Other); Lucile Packard Children's Hospital (Other); St. Jude Children's Research Hospital (Other); Seattle Children's Hospital (Other); Patient-Centered Outcomes Research Institute (Other); Alfred I. duPont Hospital for Children (Other); Children's Hospital Colorado (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 15-012103
Record Dates: First submitted 2016-05-16; First posted 2016-05-19 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Pediatric Acute Myeloid Leukemia
Keywords: Pediatric; Acute Myeloid Leukemia; Quality of Life; Neutropenia Management; Patient Centered Outcomes; Chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early Discharge Patients: Patients receiving or having received chemotherapy for AML who are discharged to outpatient management within 3 days after chemotherapy completion. Subjects will complete a health related quality of life (HRQOL) survey at baseline and again at the start of the next treatment course. Survey questions will collect information such as patient race and educational level.
- Inpatient Management Patients: Patients receiving or having received chemotherapy for AML who remain in the hospital more than 3 days after chemotherapy completion. Subjects will complete a health related quality of life (HRQOL) survey at baseline and again at the start of the next treatment course. Survey questions will collect information such as patient race and educational level.

SUMMARY:
Treatment for pediatric acute myeloid leukemia (AML) involves intensive chemotherapy regimens that result in periods of profound neutropenia leaving patients susceptible to severe infectious complications. Infectious complications are the leading cause of treatment related mortality among AML patients, but there are little clinical data to inform whether management of neutropenia post AML chemotherapy should occur in an outpatient or inpatient setting. Further, no studies have been conducted that assess the impact of neutropenia management strategy on the quality of life of pediatric patients with AML and their caregivers.

DETAILED DESCRIPTION:
This is a prospective observational cohort study, where the primary objective of this study is to compare patient and caregiver quality of life and other patient-centered outcomes for inpatient versus outpatient management of neutropenia in children with AML or MDS receiving standard intensive AML frontline chemotherapy.

Local study investigators (pediatric oncologists and study coordinators) at each of the fifteen participating pediatric institutions will communicate on a weekly basis with their inpatient leukemia service to identify AML or MDS patients potentially eligible for study enrollment. Once identified, study personnel will review each patient for study eligibility criteria. Three visits with the patient and their caregivers will occur: a screening visit, initial survey visit, and a follow-up visit.

Screening Visit: The eligibility criteria for participation will be confirmed prior to approaching for consent. Eligible patients interested in the study will be approached for consent at any time from AML/MDS diagnosis through last day of chemotherapy in the treatment course under study. In some cases, the patient's caregivers may not be present in the hospital to provide consent. In these cases, study personnel will obtain verbal consent from the caregivers and child assent (if appropriate).

Visit 1 will occur prior to the last day of chemotherapy administration in the course. This visit will include:

* 2 Brief demographic surveys to capture covariates unavailable in the medical record
* Baseline health-related quality of life (HRQOL) surveys
* A baseline financial toxicity assessment

Surveys will be administered via paper or a smart device and will last a total of 15-30 minutes per respondent. In the case that the child is 5 years of age or older, the child self-report and parent proxy-report scales will be separately administered to the child and caregiver, respectively. If the child is under 5 years of age, only the parent-proxy version will be administered. Only the caregiver completes the baseline financial toxicity assessment. We will provide a $25 gift card to each child-parent dyad upon completion of the baseline surveys

Visit 2 will occur within the period after absolute neutrophil count recovery and ideally prior to the start of the subsequent course of chemotherapy, but no later than the last day of chemotherapy in that next treatment course. This visit will include:

* Follow-up HRQOL surveys
* Patient-centered outcome survey developed previously from qualitative interviews of AML patients and their caregivers
* A follow-up financial toxicity assessment

Surveys will be administered via paper or a smart device and will last a total of 15-30 minutes per respondent. In the case that the child is 5 years of age or older, the child self-report and parent proxy-report scales will be administered to the child and caregiver, respectively. If the child is under 5 years of age, only the parent-proxy version will be administered. The follow-up financial toxicity assessment and the patient-centered outcome survey are completed by the caregiver only. We will provide a $25 gift card to each child-parent dyad upon completion of the follow-up surveys.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be enrolled as patient-caregiver dyads. The patient must be:

   * Less than 19 years of age at diagnosis.
   * Patient is English or Spanish literate.
   * Receiving chemotherapy for AML between June 1, 2016 and December 31, 2019.
2. Participants will be enrolled as patient-caregiver dyads. The caregiver must be:

   * English or Spanish literate.
   * The legal guardian of a patient receiving chemotherapy for AML between June 1, 2016 and December 31, 2019.
3. Parental/caregiver informed consent and, if appropriate, child assent.

Exclusion Criteria:

1. Patients being treated for relapsed AML
2. Patients with Acute Promyelocytic Leukemia (APML)
3. Patients undergoing stem cell transplant (SCT)
4. Patients receiving reduced intensity frontline chemotherapy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include all AML patients who are receiving a planned chemotherapy course at any of the fifteen pediatric institutions across the US between June 1, 2016 and December 31, 2019. Patients discharged within 3 days after chemotherapy completion will be categorized as 'early discharge' to outpatient management during neutropenia. Patients remaining in the hospital more than 3 days after chemotherapy completion will be categorized as inpatient management.
  Caregivers of these patients will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2016-09; Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aplenc, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (15):
- United States (15):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Nemours/Alfred I DuPont Hospital for Children, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute/Boston Children's Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
only aggregate and de-identified data will be shared upon appropriate request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Discharge Patients: Patients receiving or having received chemotherapy for AML who are discharged to outpatient management within 3 days after chemotherapy completion. Subjects will complete a health related quality of life (HRQOL) survey at baseline and again at the start of the next treatment course. Survey questions will collect information such as patient race and educational level.
  HRQOL questions will be scored on a 5-point Likert response scale (0=never a problem to 4=almost always a problem). The total score includes a 23 item multidimensional core (physical, emotional, social and school functioning); an 18 item multidimensional fatigue scale (general, sleep/rest and cognitive fatigue) and a 27 item multidimensional cancer module (pain, nausea, anxiety, communication, and cognitive problems). Total score is calculated with a lower score representing a higher health related quality of life.
- Inpatient Management Patients: Patients receiving or having received chemotherapy for AML who remain in the hospital more than 3 days after chemotherapy completion. Subjects will complete a health related quality of life (HRQOL) survey at baseline and again at the start of the next treatment course. Survey questions will collect information such as patient race and educational level.
  HRQOL questions will be scored on a 5-point Likert response scale (0=never a problem to 4=almost always a problem). The total score includes a 23 item multidimensional core (physical, emotional, social and school functioning); an 18 item multidimensional fatigue scale (general, sleep/rest and cognitive fatigue) and a 27 item multidimensional cancer module (pain, nausea, anxiety, communication, and cognitive problems). Total score is calculated with a lower score representing a higher health related quality of life.
Period: Overall Study
Arm/Group | Early Discharge Patients | Inpatient Management Patients
Started (366 patients were screened for eligibility for Aim 3. 154 patients consented for Aim 3.) | 60 | 94
Completed | 43 | 77
Not Completed | 17 | 17

BASELINE CHARACTERISTICS:
Population: Of the 154 consented patients, only 97 were discharge eligible or within the analyzed population, thus only 97 patients were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Discharge Patients | Inpatient Management Patients | Total
Number analyzed (Participants) | 22 | 75 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 75 | 97
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 38 | 46
  Male | 14 | 37 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 10 | 56 | 66
  Race: Black | 5 | 6 | 11
  Race: Asian | 2 | 5 | 7
  Race: Other | 5 | 6 | 11
  Race: Not recorded in EMR | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Ethnicity: Hispanic Ethnicity | 4 | 13 | 17
  Hispanic Ethnicity: Not Hispanic Ethnicity | 18 | 62 | 80
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 75 | 97

OUTCOME MEASURES:

1. Primary Outcome: Compare Differences in HRQOL Scores Between Outpatient Versus Inpatient Management
Description: 1 Course of Chemotherapy (Approximately 30-40 days). The primary outcome of interest was patient health-related quality of life (HRQOL) measured using the acute PedsQL™ 4.0 Generic Core Scales.31 These scales use a 7-day time frame. The multidimensional assessment includes items in four domains: physical functioning, emotional functioning, social functioning, and school functioning. Respondents document responses to each question using a 5-point Likert scale anchored by never a problem (0) to almost always a problem (4). PedsQL™ items were reverse scored and linearly transformed to a scale of 0 to 100 such that higher scores reflect better HRQOL.
Time Frame: PedsQL assessments were administered at two points - at the start of the study-contributed chemotherapy course prior to the patient becoming neutropenic (baseline) and again within the period between neutropenia resolution (follow-up); follow-up reported.
Population: Participants who completed evaluable PedsQL follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Discharge Patients | Inpatient Management Patients
Number analyzed (Participants) | 22 | 75
score on a scale | 70.1 (18.9) | 68.7 (19.4)

2. Secondary Outcome: Responses From Structured Patient-centered Outcome Surveys
Description: Information from semi-structured patient outcome surveys completed by patients and caregivers will be collected to evaluate the relationship between neutropenia management strategy (inpatient versus outpatient) and outcomes reported by patients and caregivers.
Time Frame: 1 Course of Chemotherapy (Approximately 30-40 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored for the duration of the study because there was no study intervention.
Description: There was no study intervention, only survey administration and collection.
Arm/Group | Early Discharge Patients | Inpatient Management Patients
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT02777021/Prot_SAP_000.pdf